CLINICAL TRIAL: NCT05714956
Title: Understanding the Needs of Parents and Providers With Mothers and Babies Online (eMB): A User Centered Approach
Brief Title: Pilot Study of Mothers and Babies Online in Home Visiting
Acronym: eMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Palo Alto University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Darius Tandon, Director, Institute for Public Health and Medicine (IPHAM) - Center for Community Health; Associate Professor of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00216763; 5P50MH119029-03 (NIH)
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Perinatal Depression
Keywords: eHealth; Home Visiting; perinatal; depression; perinatal depression; user centered design; digital mental health
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): eMB consists of 8 sessions that correspond with key cognitive-behavioral therapy (CBT) elements: pleasant activities, thoughts, and social support/contact with others. Integrated throughout eMB are activities and skills based on attachment theory that emphasize how each CBT module relates to promoting a strong, nurturing connection between parent and child. eMB includes informational pages, short audio/video clips, images of infants and pregnant women, and worksheets for participants to enter personalized information in response to the lesson content. eMB is individually guided without facilitation, b) clients control the pace by which they review online content, c) and clients can review online content as many times as they like. Participants who receive eMB will also complete assessments at baseline, 1 week post-intervention, and 3 months post-intervention.
  Interventions: Behavioral: Mothers and Babies Online (eMB)
- Home Visiting Usual Care (No Intervention): Core content of home visiting program services typically address: (a) preparation for childbirth and having a young child in the home, (b) provision of emotional and tangible [e.g., diapers, formula] support, (c) discussion of infant and young child development, (d) linkages to prenatal and pediatric care, and (e) referrals to community resources for social and health services. Those receiving usual care home visiting will not receive any eMB or MB course content. Once study participation is completed, the home visitor may introduce eMB to the participant if they are interested. Participants in the control group will also complete assessments at baseline, 1 week post-intervention (i.e., following 8 weeks of usual home visiting services), and 3 months post-intervention (i.e.g, following 8 weeks of usual home visiting services).

INTERVENTIONS:
Behavioral: Mothers and Babies Online (eMB) — This study's intervention is called Mothers and Babies Online or "eMB", which consists of 8 sessions that correspond with key cognitive-behavioral therapy (CBT) elements: pleasant activities, thoughts, and social support/contact with others. Integrated throughout eMB are activities and skills based on attachment theory that emphasize how each CBT module relates to promoting a strong, nurturing connection between parent and child. eMB includes informational pages, short audio/video clips, images of infants and pregnant women, and worksheets for participants to enter personalized information in response to the lesson content. eMB is individually guided without facilitation, b) clients control the pace by which they review online content, c) and clients can review online content as many times as they like. Participants who receive eMB will also complete assessments at baseline, 1 week post-intervention, and 3 months post-intervention.
  Arms: Intervention

SUMMARY:
The investigators propose a pilot randomized controlled trial (RCT) that examines how the redesigned version of Mothers and Babies Online (eMB) can be delivered in the context of home visiting (HV) programs that serve pregnant individuals and new mothers across the United States. The PI, Dr. Darius Tandon (Northwestern University), has conducted extensive research on the in-person Mothers and Babies (MB) intervention with HV programs and has received interest from one of the largest HV models-Parents as Teachers (PAT)-to explore the use of eMB with pregnant individuals that they serve.

DETAILED DESCRIPTION:
This pilot study examining how to incorporate Mothers and Babies Online or "eMB" into home visiting program workflows will have three Specific Aims:

1. Employ a user-centered design (UCD) approach in which investigators will conduct semi-structured qualitative interviews with key home visiting stakeholders (n = 10 parent clients, n = 5 home visitors) to generate recommendations on a) how to integrate eMB into home visiting program workflows, b) appropriate strategies for home visitors providing human support to support eMB engagement, c) reactions to the messaging and tone of eMB; and c) potential barriers and facilitators to eMB engagement.
2. Conduct a small randomized trial that examines the feasibility, acceptability, and effectiveness of eMB when implemented in home visiting programs. Investigators will recruit 50 pregnant individuals and new mothers from 5-8 Parents as Teachers programs that serve rural communities. Investigators have chosen to focus on rural communities given the challenges associated with in-person intervention delivery in those settings. These individuals will be randomized where 40 individuals will complete the eMB intervention and 10 will serve as controls receiving usual HV services. Participants who are at-risk for developing postpartum depression will be eligible for the study. Investigators will assess risk for postpartum depression using two screening tools-the Edinburgh Postnatal Depression Scale (EPDS) and the Postpartum Depression Predictors Inventory (PDPI). Women scoring in the mild/moderate range (5-14) on the EPDS or scoring >3.5 on the PDPI are considered at elevated risk for postpartum depression. Data from the UCD phase will be used to develop study protocols for implementing eMB, including how home visitors providing human support/coaching while clients are engaged with eMB. Investigators will collect maternal self-report data on depressive symptoms, perceived stress, and other mental health outcomes at baseline (pre-intervention), 1-week post-intervention, and 3-months post-intervention.
3. Conduct brief semi-structured interviews with n = 15 parent clients who received eMB during the pilot RCT and n = 5 home visitors who provided eMB coaching during the pilot RCT to understand user experience with eMB (with particular emphasis on understanding any human support/coaching component), which will guide any necessary modifications to the intervention protocol. Investigators will also conduct brief semi-structured interviews with program managers from participating Parents as Teachers (PAT) programs and PAT leadership to assess organizational-level barriers and facilitators to eMB uptake, which will inform future research directions related to the implementation of eMB.

ELIGIBILITY:
Inclusion Criteria:

1. Are enrolled in home visiting services
2. Are 16 years or older
3. Are English Proficient (reading, speaking, and writing)
4. Are currently pregnant or have a young child up to 6 months
5. Have internet access
6. Have access to an electronic device (cell phone, laptop, tablet, etc.)
7. Are at risk for developing perinatal depression as defined by one or more of the following: a score of 5-14 on the Edinburgh Postnatal Depression Scale (EPDS), a score of >3.5 on the Postpartum Depression Predictors Inventory (PDPI), personal history of depression, and/or familial history of depression.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | T1 (prior to starting intervention), T2 (1 week post-intervention), T3 (3 months post-intervention)
  Depression will be assessed using the Center for Epidemiological Studies-Depression Scale, which is a 20-item measure that asks participants to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Scores range from 0-60 with higher scores indicating greater depressive symptomatology

SECONDARY OUTCOMES:
Change in perceived stress | T1 (prior to starting intervention), T2 (1 week post-intervention), T3 (3 months post-intervention)
  Perceived stress will be assessed using the 10-item Perceived Stress Scale (PSS-10), which asks respondents to indicate their levels of perceived stress in the last month, with a response of "0" indicating "Never" and a response of "4" indicating "very often."
Change in anxiety symptoms | T1 (prior to starting intervention), T2 (1 week post-intervention), T3 (3 months post-intervention)
  Symptoms of anxiety will be measured using the Generalized Anxiety Disorder-7, which is a 7-item measure that aligns with the Diagnostic and Statistical manual of Mental Disorders (DSM-5) criteria for GAD and assesses anxiety symptom frequency and severity. This instrument has scores ranging from 0-21 with higher scores indicating greater anxiety symptoms.
Change in parenting sense of competence | T1 (prior to starting intervention), T2 (1 week post-intervention), T3 (3 months post-intervention)
  Parenting sense of competence (PSOC) is a 17-item scale developed to assess parenting self-esteem. The scale includes two rationally derived scales, Skill-Knowledge and Value-Comforting, referred to as Efficacy and Satisfaction. Each item is answered on a 6-point scale ranging from strongly disagree (6) to strongly agree (1).
Chang in dimensions of couple relationships | T1 (prior to starting intervention), T2 (1 week post-intervention), T3 (3 months post-intervention)
  Dimensions of couple relationships will be measured using the Revised Dyadic Adjustment Scale , a report questionnaire that assesses seven dimensions of couple relationships within three overarching categories including consensus in decision making, values and affection, satisfaction in the relationship with respect to stability and conflict regulation, and cohesion. Scores range from 0-69 with higher scores indicating stronger relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Darius Tandon, PhD, Principal Investigator — Northwestern University
Locations (6):
- United States (6):
  - Metropolitan Family Services, Chicago, Illinois
  - Easter Seals, Joliet, Illinois
  - South Central Iowa Community Action Program, Chariton, Iowa
  - Children & Family Resource Center, Hendersonville, North Carolina
  - Carolina Health Centers, Greenwood, South Carolina
  - Newport News, Newport News, Virginia

REFERENCES:
- [Background] Evans J, Heron J, Francomb H, Oke S, Golding J. Cohort study of depressed mood during pregnancy and after childbirth. BMJ. 2001 Aug 4;323(7307):257-60. doi: 10.1136/bmj.323.7307.257. PMID 11485953
- [Background] Gaynes BN, Gavin N, Meltzer-Brody S, Lohr KN, Swinson T, Gartlehner G, Brody S, Miller WC. Perinatal depression: prevalence, screening accuracy, and screening outcomes. Evid Rep Technol Assess (Summ). 2005 Feb;(119):1-8. doi: 10.1037/e439372005-001. No abstract available. PMID 15760246
- [Background] Moses-Kolko EL, Roth EK. Antepartum and postpartum depression: healthy mom, healthy baby. J Am Med Womens Assoc (1972). 2004 Summer;59(3):181-91. PMID 15354371
- [Background] Segre LS, O'Hara MW, Arndt S, Stuart S. The prevalence of postpartum depression: the relative significance of three social status indices. Soc Psychiatry Psychiatr Epidemiol. 2007 Apr;42(4):316-21. doi: 10.1007/s00127-007-0168-1. Epub 2007 Feb 13. PMID 17370048
- [Background] Robertson E, Grace S, Wallington T, Stewart DE. Antenatal risk factors for postpartum depression: a synthesis of recent literature. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):289-95. doi: 10.1016/j.genhosppsych.2004.02.006. PMID 15234824
- [Background] Beebe B, Jaffe J, Buck K, Chen H, Cohen P, Blatt S, Kaminer T, Feldstein S, Andrews H. Six-week postpartum maternal self-criticism and dependency and 4-month mother-infant self- and interactive contingencies. Dev Psychol. 2007 Nov;43(6):1360-76. doi: 10.1037/0012-1649.43.6.1360. PMID 18020817
- [Background] Murray L, Cooper PJ, Wilson A, Romaniuk H. Controlled trial of the short- and long-term effect of psychological treatment of post-partum depression: 2. Impact on the mother-child relationship and child outcome. Br J Psychiatry. 2003 May;182:420-7. PMID 12724245
- [Background] National Research Council (US) and Institute of Medicine (US) Committee on the Prevention of Mental Disorders and Substance Abuse Among Children, Youth, and Young Adults: Research Advances and Promising Interventions; O'Connell ME, Boat T, Warner KE, editors. Preventing Mental, Emotional, and Behavioral Disorders Among Young People: Progress and Possibilities. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32775/ PMID 20662125
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders: DSM-5. ManMag; 2003.
- [Background] Howell EA, Mora PA, Horowitz CR, Leventhal H. Racial and ethnic differences in factors associated with early postpartum depressive symptoms. Obstet Gynecol. 2005 Jun;105(6):1442-50. doi: 10.1097/01.AOG.0000164050.34126.37. PMID 15932842
- [Background] Mora PA, Bennett IM, Elo IT, Mathew L, Coyne JC, Culhane JF. Distinct trajectories of perinatal depressive symptomatology: evidence from growth mixture modeling. Am J Epidemiol. 2009 Jan 1;169(1):24-32. doi: 10.1093/aje/kwn283. Epub 2008 Nov 10. PMID 19001135
- [Background] Bennett HA, Einarson A, Taddio A, Koren G, Einarson TR. Prevalence of depression during pregnancy: systematic review. Obstet Gynecol. 2004 Apr;103(4):698-709. doi: 10.1097/01.AOG.0000116689.75396.5f. PMID 15051562
- [Background] Dolbier CL, Rush TE, Sahadeo LS, Shaffer ML, Thorp J; Community Child Health Network Investigators. Relationships of race and socioeconomic status to postpartum depressive symptoms in rural African American and non-Hispanic white women. Matern Child Health J. 2013 Sep;17(7):1277-87. doi: 10.1007/s10995-012-1123-7. PMID 22961387
- [Background] Holzman C, Eyster J, Tiedje LB, Roman LA, Seagull E, Rahbar MH. A life course perspective on depressive symptoms in mid-pregnancy. Matern Child Health J. 2006 Mar;10(2):127-38. doi: 10.1007/s10995-005-0044-0. Epub 2006 Jan 7. PMID 16400535
- [Background] Schmit S, Schott L, Pavetti L, Matthews H. Effective, Evidence-Based Home Visiting Programs in Every State at Risk if Congress Does Not Extend Funding. 2015;http://www.cbpp.org/research/effective-evidence-based-home-visiting-programs-in-every-state-at-risk-if-congress-does-not. Accessed February 10, 2016.
- [Background] Avellar S, Paulsell D, Sama-Miller E, Grosso PD, Akers L, Kleinman R. Home visiting evidence of effectiveness review: Executive summary. Mathematica Policy Research;2013.
- [Background] U.S. Department of Health and Human Services, Administration for Children and Families, Office of Planning and Evaluation. Depression in the Lives of Early Head Start Families: Research to Practice Brief. 2006; http://www.acf.hhs.gov/programs/opre/resource/depression-in-the-lives-of-early-head-start-families-research-to-practice. Accessed January 15, 2014. Accessed January 15, 2016.
- [Background] U.S. Department of Health and Human Services, Health Resources and Services Administration, Maternal and Child Health Bureau. A Comprehensive Approach for Community-Based Programs to Address Intimate Partner Violence and Perinatal Depression. 2013; http://mchb.hrsa.gov/pregnancyandbeyond/depression/partnerviolence/partnerviolenceandperinataldepression.pdf.Accessed February 10 2016.
- [Background] Prevent Child Abuse America. Healthy Families America Critical Elements. 2001; http://www.healthyfamiliesamerica.org/downloads/critical_elements_rationale.pdf. Accessed January 15, 2016.
- [Background] Ammerman RT, Putnam FW, Bosse NR, Teeters AR, Van Ginkel JB. Maternal Depression in Home Visitation: A Systematic Review. Aggress Violent Behav. 2010 May;15(3):191-200. doi: 10.1016/j.avb.2009.12.002. PMID 20401324
- [Background] Ammerman RT, Putnam FW, Altaye M, Chen L, Holleb LJ, Stevens J, Short JA, Van Ginkel JB. Changes in depressive symptoms in first time mothers in home visitation. Child Abuse Negl. 2009 Mar;33(3):127-38. doi: 10.1016/j.chiabu.2008.09.005. Epub 2009 Mar 27. PMID 19328548
- [Background] Chazan-Cohen R, Ayoub C, Pan BA, Roggman L, Raikes H, Mckelvey L, Whiteside-Mansell L, Hart A. It takes time: Impacts of Early Head Start that lead to reductions in maternal depression two years later. Infant Ment Health J. 2007 Mar;28(2):151-170. doi: 10.1002/imhj.20127. PMID 28640556
- [Background] Tandon SD, Parillo KM, Jenkins C, Duggan AK. Formative evaluation of home visitors' role in addressing poor mental health, domestic violence, and substance abuse among low-income pregnant and parenting women. Matern Child Health J. 2005 Sep;9(3):273-83. doi: 10.1007/s10995-005-0012-8. PMID 16240078
- [Background] McFarlane E, Burrell L, Duggan A, Tandon D. Outcomes of a Randomized Trial of a Cognitive Behavioral Enhancement to Address Maternal Distress in Home Visited Mothers. Matern Child Health J. 2017 Mar;21(3):475-484. doi: 10.1007/s10995-016-2125-7. PMID 27535131
- [Background] Tandon SD, Leis JA, Mendelson T, Perry DF, Kemp K. Six-month outcomes from a randomized controlled trial to prevent perinatal depression in low-income home visiting clients. Matern Child Health J. 2014 May;18(4):873-81. doi: 10.1007/s10995-013-1313-y. PMID 23793487
- [Background] Tandon SD, Ward EA, Hamil JL, Jimenez C, Carter M. Perinatal depression prevention through home visitation: a cluster randomized trial of mothers and babies 1-on-1. J Behav Med. 2018 Oct;41(5):641-652. doi: 10.1007/s10865-018-9934-7. Epub 2018 May 15. PMID 29766470
- [Background] US Preventive Services Task Force; Curry SJ, Krist AH, Owens DK, Barry MJ, Caughey AB, Davidson KW, Doubeni CA, Epling JW Jr, Grossman DC, Kemper AR, Kubik M, Landefeld CS, Mangione CM, Silverstein M, Simon MA, Tseng CW, Wong JB. Interventions to Prevent Perinatal Depression: US Preventive Services Task Force Recommendation Statement. JAMA. 2019 Feb 12;321(6):580-587. doi: 10.1001/jama.2019.0007. PMID 30747971
- [Background] McCurdie T, Taneva S, Casselman M, Yeung M, McDaniel C, Ho W, Cafazzo J. mHealth consumer apps: the case for user-centered design. Biomed Instrum Technol. 2012 Fall;Suppl:49-56. doi: 10.2345/0899-8205-46.s2.49. No abstract available. PMID 23039777
- [Background] Lyon AR, Koerner K. User-Centered Design for Psychosocial Intervention Development and Implementation. Clin Psychol (New York). 2016 Jun;23(2):180-200. doi: 10.1111/cpsp.12154. Epub 2016 Jun 17. PMID 29456295
- [Background] Virzi, R.A., J.F. Sorce, and L.B. Herbert. A comparison of three usability evaluation methods: Heuristic, think-aloud, and performance testing. in Human Factors and Ergonomics Society Annual Meeting. 1993. Los Angeles, CA: Sage Publications.
- [Background] Bradley EH, Curry LA, Devers KJ. Qualitative data analysis for health services research: developing taxonomy, themes, and theory. Health Serv Res. 2007 Aug;42(4):1758-72. doi: 10.1111/j.1475-6773.2006.00684.x. PMID 17286625
- [Background] Fusch, P.I. and L.R. Ness, Are we there yet? Data saturation in qualitative research. Qualitative Report, 2015. 20(9): p. 1408-1416.
- [Background] Guest, G., A. Bunce, and L. Johnson, How many interviews are enough? An experiment with data saturation and variability. Field Methods, 2006. 18(1): p. 59-82.
- [Background] Faulkner L. Beyond the five-user assumption: benefits of increased sample sizes in usability testing. Behav Res Methods Instrum Comput. 2003 Aug;35(3):379-83. doi: 10.3758/bf03195514. PMID 14587545
- [Background] DeSantis L, Ugarriza DN. The concept of theme as used in qualitative nursing research. West J Nurs Res. 2000 Apr;22(3):351-72. doi: 10.1177/019394590002200308. PMID 10804897
- [Background] Hill, C.E., et al., Consensual qualitative research: An update. Journal of counseling psychology, 2005. 52(2): p. 196.
- [Background] Hill, C.E., B.J. Thompson, and E.N. Williams, A guide to conducting consensual qualitative research. The Counseling Psychologist, 1997. 25(4): p. 517-572.